CLINICAL TRIAL: NCT05154071
Title: Impact of the Implementation of a Referral Veno-venous Extracorporeal Membrane Oxygenation Centre on Mortality
Acronym: ECMO UNIT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: NGUYEN 2021-3
Record Dates: First submitted 2021-10-21; First posted 2021-12-10 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECMO VV dedicated unit: Patient having benefited from an ECMO within the structured care unit
  Interventions: Other: Collection of medical data
- ECMO VV without dedicated unit: Patient having benefited from an ECMO without the structured care unit
  Interventions: Other: Collection of medical data

INTERVENTIONS:
Other: Collection of medical data — Collection of adverse events, of mortality, length of hospitalization

SUMMARY:
Current evidence suggest that regrouping patient supported by veno-venous ECMO in high-volume centre could improve outcome. A dedicated ECMO unit was implemented in Dijon.

The objective of the present study was to evaluate the implementation of this unit. The hypothesis was that patient taken care within this structured care system would have lower mortality.

This research comprises a retrospective observational study conducted in Dijon university hospital

ELIGIBILITY:
Inclusion Criteria:

* patient in an adult Dijon ICUs supported by veno-venous ECMO
* patient hospitalized between January the 1st 2011 and June the 30th 2021

Exclusion Criteria:

* Refusal to participate,
* patient admitted to pediatric ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients supported by veno-venous ECMO
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 90 days

SECONDARY OUTCOMES:
Rate of ECMO adverse events | through study completion, an average of 3 years
Hospital length of stay | through study completion, an average of 3 years
ICU length of stay | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Nguyen M, Kabbout V, Berthoud V, Gounot I, Dransart-Raye O, Douguet C, Bouchot O, Morgant MC, Bouhemad B, Guinot PG. Implementation of a regional multidisciplinary veno-venous extracorporeal membrane oxygenation unit improved survival: a historical cohort study. Can J Anaesth. 2022 Jul;69(7):859-867. doi: 10.1007/s12630-022-02259-4. Epub 2022 May 2. PMID 35501590